CLINICAL TRIAL: NCT06200194
Title: Early Intervention for Premyopic Children: A Comparison Study of Defocus Integrated Multiple Segments Spectacle Lenses, 0.01% Atropine and Usual Care for Myopia Prevention
Brief Title: Early Intervention for Premyopic Children
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Principal Investigator, Der-Chong Tsai, MD PhD, Principal Investigator, National Yang Ming Chiao Tung University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NYCUH2023A018
Record Dates: First submitted 2023-12-28; First posted 2024-01-10 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Myopia; Preschool
MeSH Terms: conditions — Myopia | interventions — Atropine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- DIMS lens (Experimental): DIMS spectacle lenses. Daily wear for 1.5 years.
  Interventions: Device: MiyoSmart Spectacles
- 0.01% Atropine (Experimental): 0.01% Atropine. One drop per eye, per day, for 1.5 years.
  Interventions: Drug: 0.01% atropine
- Usual care (No Intervention): Usual care including promoting outdoor time

INTERVENTIONS:
Device: MiyoSmart Spectacles — No power in the central optic zone of DIMS lens for premyopic children with normal vision. Before entering elementary school, eligible preschoolers are asked to wear the DIMS spectacles after kindergarten hours and during weekends and holidays. After entering elementary school, full-time mode wearing of DIMS spectacles is required.
  Other Names: MiyoSmart (Hoya, Tokyo, Japan)
  Arms: DIMS lens
Drug: 0.01% atropine — daily use of non-preservative 0.01% atropine eye drop for each eye over the study period.
  Other Names: "AIM" Atropine Eye Drops 0.01% (AIMedicine, Taipei, Taiwan)
  Arms: 0.01% Atropine

SUMMARY:
The purpose of this research project is to add evidence of pharmacological (0.01% atropine) and optical (Defocus Integrated Multiple Segments spectacle lenses) approaches for myopia prevention among premyopic preschoolers, which may contribute to a better understanding of the intervention strategy for myopia control in premyopic children.

DETAILED DESCRIPTION:
With more popularity of screen-based digital devices in the post-pandemic era, childhood myopia prevention and control has encountered a tough challenge on a global scale. Though the protective effect of spending more time outdoors has been well proven, the optimal practice for preventing or delaying the early onset of childhood myopia still needs further investigations, particularly in pre-myopic children around the school entrance age. It has been reported that there is a double-digit increase in myopia prevalence before and after elementary school entry, and young children with early-onset myopia are at great risk of rapid progression to high myopia later in life. Most recently, nightly use of 0.05% atropine eye drops is effective in reducing the incidence of childhood myopia. However, photophobia is a common adverse effect of higher concentration atropine, which may hinder children from daytime outdoor activities. Besides, little is known about the optical approach for myopia prevention in the existing literature. These unmet demands in clinical practice motivate us to propose a randomized controlled trial on myopia prevention with optical (Defocus Incorporated Multiple Segments [DIMS] spectacle lenses) or pharmacological (0.01% atropine eye drops) modalities among pre-myopic preschoolers aged 5-6 years. To explore the adaptability and feasibility of DIMS spectacle lenses for pre-myopic children with normal visual acuity, we have conducted a pilot study and revealed that all 24 subjects can tolerate daily full-time wearing of DIMS spectacle lenses without significant visual complaints. In this proposal, we plan to recruit a total of 234 eligible participants who have been identified as pre-myopic and asymptomatic in a population-based eye care program in Yilan County. Eligible subjects will be randomly assigned to the DIMS spectacles (n=78), 0.01% atropine (n=78), and usual care (n=78) groups. Less environmental pressure is hypothesized in preschool compared with elementary school. Hence, pre-myopic children will be asked to wear DIMS spectacle lenses in a stepwise pattern: at-home wearing in the preschool stage and full-time in the elementary school stage. Cycloplegic spherical equivalent (SE) refraction and axial length will be measured every 3 months over the 18-month follow-up period. The primary outcome is the changes in mean cycloplegic SE over the study period in each group. The secondary outcomes include the cumulative percentage of incident myopia, the cumulative percentage of a fast myopic shift of SE, and the changes in mean axial length over the study period in each group. This proposed project may offer insight into the intervention strategy for myopia prevention and evoke the possibility of a reinvented eye care policy that may focus on early identification and intervention for pre-myopic preschoolers.

ELIGIBILITY:
Inclusion Criteria:

* Age at enrollment: 5-6 years old (the senior grade of kindergarten)
* Cycloplegic SE of the eye with less SE (less positive or more negative refractive error): < +1.00 D and > -0.50 D
* Astigmatism: 1.0 D or less in both eyes
* Anisometropia: 1.50 D or less
* Monocular uncorrected visual acuity: 6/7.5 or better in both eyes
* Either of the parents with moderate myopia
* Acceptance of random group allocation
* Submission of complete informed consent.

Exclusion Criteria:

* Strabismus or any ocular motility disorder
* Any ophthalmic and systemic disorders that might affect visual functions or refractive development
* Previous treatment of atropine or other myopia control intervention

Ages: 5 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 240 (Estimated)
Dates: Start 2024-10-06 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Myopic shift of spherical equivalent refraction | 18 months
  The change of mean cycloplegic spherical equivalent refraction over 1.5 years

SECONDARY OUTCOMES:
Axial length elongation | 18 months
  The change of mean axial length over 1.5 years
Incidence of myopia | 18 months
  the cumulative percentage of incident myopia
Fast myopic shift of spherical equivalent refraction | 18 months
  the cumulative percentage of fast myopic shift of spherical equivalent refraction

CONTACTS AND LOCATIONS:
Overall Officials: Der-Chong Tsai, MD, PhD, Principal Investigator — National Yang Ming Chiao Tung University Hospital
Locations (1):
- National Yang Ming Chiao Tung University Hospital, Yilan, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yang HY, Tsai DC, Yang YC, Wang CY, Lee CW, Huang PW. Efficacy of defocus incorporated multiple segments (DIMS) lenses and low-dose atropine on retarding myopic shift among premyopic preschoolers: Protocol for a prospective, multicenter, randomized controlled trial. PLoS One. 2024 Dec 31;19(12):e0312935. doi: 10.1371/journal.pone.0312935. eCollection 2024. PMID 39739826